CLINICAL TRIAL: NCT05078086
Title: Study on the Relationship of Arterial-venous Oxygen Difference and Postoperative Complications After Cardiac Surgery.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Yan, Director of Department of Anesthesiology, The Second Affiliated Hospital, Zhejiang University School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2021-0486
Record Dates: First submitted 2021-09-27; First posted 2021-10-14 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Patient Blood Management; Cardiac Surgery; Transfusion
Keywords: arterial-venous oxygen difference; Patient blood management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgery with CPB: >18 y/o patients who undergo cardiac surgery with cardiopulmonary bypass and with a preoperative additive EuroSCORE I≥ 6
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Avoidance of unnecessary blood transfusions has always been a focus of clinical research. The rate of perioperative red blood cell transfusion in patients undergoing cardiac surgery under cardiopulmonary bypass reaches between 50-70%, and the intraoperative red blood cell transfusion rate is 30-50%. Regarding whether and when to perform a blood transfusion, it is necessary to comprehensively consider the benefits and risks brought by blood transfusion.

Previous studies on blood transfusion strategies have mainly focused on the hemoglobin threshold, but the hemoglobin level does not fully reflect the level of tissue oxygenation. Mixed venous blood oxygen saturation has been widely studied as a valuable indicator reflecting the balance of oxygen delivery and oxygen consumption. But due to the difficulty of placing a pulmonary artery floating catheter for monitoring, its clinical application is limited. Central venous oxygen saturation requires only a small collection of blood samples, which can reflect the oxygen saturation of the superior vena cava, and studies have shown that it can effectively guide the blood transfusion of patients undergoing cardiac surgery. Existing studies have shown that in critically ill patients, the use of arterial-venous oxygen difference > 3.7 mL as an indicator to guide blood transfusion can lead to a higher 90-day survival rate. However, the relationship between the arterial-venous oxygen difference and the incidence of adverse events in cardiac surgery patients under CPB remains unclear. Whether increasing the arterial-venous oxygen difference during surgery can reduce the incidence of postoperative adverse events remains to be clarified.

This study intends to collect intraoperative arterial blood and central venous blood samples from cardiac surgery patients undergoing CPB, and analyze the relationship between arterial-venous oxygen difference and the incidence of postoperative adverse events.

DETAILED DESCRIPTION:
The >18 y/o patients who undergo cardiac surgery with cardiopulmonary bypass and with a preoperative additive EuroSCORE I≥ 6 are enrolled. Blood samples will be collected through arteries and central venous at the following intraoperative time points: before CPB, during CPB, and after CPB. The observation will end by hospital discharge or 28 days after surgery, whichever came first. The follow-up will continue for one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Cardiovascular surgery patients with cardiopulmonary bypass
* Preoperative EuroSCORE I≥6（European System for Cardiac Operative Risk Evaluation)
* Obtained informed consent

Exclusion Criteria:

* Patients who cannot accept blood products
* Patients who refuse to accept transfusion
* Patients with autologous blood reserve before surgery
* Patients who are going to receive heart transplantation or have undergone heart transplantation
* Patients who have undergone ventricular assist device implantation surgery
* Patients who refuse to participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to high risk patients undergoing cardiac surgery with cardiopulmonary bypass (CPB)
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Composite outcome of mortality and serious morbidity (cardiac, renal, and neurological events) | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Composite incidence of any one of the following events occurring during the hospitalization : (1) all-cause mortality; (2) myocardial infarction; (3) new renal failure requiring dialysis; or (4) new focal neurological deficit (stroke)

SECONDARY OUTCOMES:
Incidence of any independent component of the primary outcome | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Incidence of any independent component of the primary outcome (all-cause mortality, myocardial infarction, new renal failure requiring dialysis, and new focal neurological deficit (stroke))
Blood product transfusion | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Time, category, and volume of blood product transfusion
Length of stay in ICU | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Length of stay in ICU after surgery
Total length of hospital stay after surgery | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Total length of hospital stay after surgery
Duration of mechanical ventilation after surgery | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Total length of hospital stay after surgery
Occurrence of low cardiac output after surgery | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Need for two or more inotropes for 24 hours or more, intra-aortic balloon pump postoperatively or ventricular assist device
Infection | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Infection will be defined as septic shock with positive blood cultures; pneumonia defined as autopsy diagnosis or roentgenographic infiltrate and at least two of the following three criteria: fever, leukocytosis, and positive sputum culture; and/or deep sternal or leg wound infection requiring intravenous antibiotics and/or surgical debridement
Gut infarction | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  confirmed by imaging, autopsy, or through surgical means
Acute kidney injury | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  AKI defined by the KDIGO
Seizures | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Defined as generalized or focal tonic-clonic movements consistent with seizure; or EEG demonstrating epileptiform discharges; or diagnosis of seizures by neurologist or neurosurgeon consultation
Delirium | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Based on one of the following criteria: CAM-ICU/ CAM (even on 1 occasion) or ICDSC > 3 or more than one dose of haloperidol or similar antipsychotic drug or documented delirium by neurologist or neurosurgeon or psychiatrist consultation
Encephalopathy | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  Defined as unexpected delayed awakening or severely altered mental status (unconscious despite no sedative medication for more than 5 days), or encephalopathy documented by neurologist or neurosurgeon or psychiatrist consultation
Reoperation rate | From the start of surgery until hospital discharge or postoperative day 28, whichever comes first
  The rate of reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided